CLINICAL TRIAL: NCT04711226
Title: An Open-Label Study to Evaluate the Safety, Tolerability and Efficacy of Immunomodulation With AT-1501 in Adults With Type 1 Diabetes Undergoing Islet Cell Transplant
Brief Title: Safety, Tolerability and Efficacy of Immunomodulation With AT-1501 in Islet Cell Transplantation
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Anelixis Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Organization: Eledon Pharmaceuticals (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT-1501-I203; AT-1501-I203 (Other: Anelixis)
Record Dates: First submitted 2021-01-10; First posted 2021-01-15 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes; T1D; Islet Cell Transplant; AT-1501; humanized blocking antibody to CD40L; CD40L inhibitor; monoclonal antibody; Glucose Metabolism Diseases; Diabetes Mellitus, Type 1; Endocrine System Diseases; Graft; Metabolic Diseases; Immune System Diseases; Autoimmune Diseases; Hypoglycemia; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Endocrine System Diseases; Metabolic Diseases; Immune System Diseases; Autoimmune Diseases; Hypoglycemia; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- AT-1501 Single Arm (Experimental)
  Interventions: Drug: AT-1501

INTERVENTIONS:
Drug: AT-1501 — AT-1501 IV infusion

SUMMARY:
This study will evaluate the safety, tolerability and efficacy of AT-1501 in an immunomodulation regimen in adult patients with T1D undergoing an islet cell transplant.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability and efficacy of AT-1501 in an immunomodulation regimen in adult patients with T1D undergoing an islet cell transplant. This study will also provide valuable data with respect to its potential additional uses in autoimmunity and solid organ transplant. This is a single arm open-label study and up to 6 participants will be recruited at a single center in Canada.

The objectives include:

* To assess the safety and tolerability of immunomodulation with AT-1501, in combination (AT+) with rabbit anti-thymoglobulin (ATG), etanercept and mycophenolate mofetil (MMF/EC-MPS) in adults with T1D undergoing islet cell transplant.
* To assess the efficacy of immunomodulation with AT-1501 in adults with T1D undergoing islet cell transplant.

The duration of treatment may vary from participant to participant and could be up to 20 months. Participants may receive up to 2 islet cell transplants.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18-65 years of age
2. A diagnosis of T1D ≥5 years with onset of disease at <40 years of age
3. Involvement in intensive diabetes management as directed by an endocrinologist or diabetologist with at least 3 clinical evaluations within the 12 months prior to Screening; using an insulin pump or multiple daily injection (MDI) insulin therapy; and, unable to achieve acceptable metabolic control because of the occurrence of severe hypoglycemia
4. At least 2 unexplained SHEs not secondary to a missed meal or dosing error, etc., in the 12 months prior to Screening
5. Glycosylated hemoglobin (HbA1c) level greater than 7% (53 mmol/mol) and less than 9.5% (80 mmol/mol) inclusive
6. Absence of stimulated C peptide (< 0.3 ng/mL) in response to a mixed meal tolerance test (MMTT) measured at 60 and 90 minutes after the start of consumption
7. Reduced awareness of hypoglycemia as defined by a Clarke Score [Clarke 1995] of 4 or more at the time of Screening, during the Screening period and within the last 6 months prior to the transplant

Exclusion Criteria:

1. Any previous transplant
2. HbA1c level less than 7% (53 mmol/mol)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Safety- Adverse Events (AE) and Adverse Events of Special Interest (AEoSI) | Accessed from date of transplant through 1 year post transplant for approximately 2 years
  Incidence of adverse events
Efficacy- Insulin independence | Days 75 , Day 365 post-first transplant, and final transplant and 1 year after discontinuation of AT-1501
  Change in the proportion of participants that become insulin independent at Days 75 and 365 post-first, and final transplant

SECONDARY OUTCOMES:
Efficacy- Graft failure | Day 365
  Proportion of participants with graft failure
Efficacy- Durability of insulin independence- long term | 2 and 3 years after discontinuation of AT- 1501
  Change in the proportion of participants that become insulin independent at year 2 and year 3
Efficacy- HbA1c | Day 365 and free of serious hypoglycemic events from Day 28 to 365 post-first transplant
  * Proportion of participants with HbA1c <7.0% (53 mmol/mol) and free of serious hypoglycemic events (SHEs)
  * Proportion of participants with HbA1c ≤6.5% (48 mmol/mol) and free from SHEs

OTHER OUTCOMES:
Exploratory- Hypoglycemia unawareness (using the method of Clarke) | Day 75, 365, and 1, 2 and 3 years after discontinuation of AT-1501
  Proportion of participants with hypoglycemia unawareness
Exploratory- Glycemic lability (using CGMS) | Day 75, 365, and 1, 2 and 3 years after discontinuation of AT-1501
  Change in glycemic lability using CGMS- Continuous Glucose Monitoring System
Exploratory- Glycemic variability (using CGMS) | Day 75, 365, and 1, 2 and 3 years after discontinuation of AT-1501
  Change in glycemic variability using CGMS- Continuous Glucose Monitoring System
Exploratory- Albumin excretion ratio (AER) | Day 365 post-first, and final transplant
  Change in albumin excretion ratio (AER)
Exploratory- eGRF | Day 365 post-first, and final transplant
  Change in eGRF
Exploratory- Macroalbuminemia | Day 365 post-first, and final transplant
  Change in percent new macroalbuminemia
Exploratory- biomarkers of tissue damage and inflammation | Day -2, 3, 14, 28, 75, 175, 364
  Biomarkers
Exploratory -Pharmacokinetic Parameters-AUC | T=0 (pre infusion), 1 (end of infusion), 2, 4, 8, 12, 24 and 48 hrs.
  Pharmacokinetics (PK) of AT-1501
Exploratory- Pharmacokinetic Parameters-Cmax | T=0 (pre infusion), 1 (end of infusion), 2, 4, 8, 12, 24 and 48 hrs.
  Pharmacokinetics (PK) of AT-1501
Exploratory- Pharmacokinetic Parameters-CL | T=0 (pre infusion), 1 (end of infusion), 2, 4, 8, 12, 24 and 48 hrs.
  Pharmacokinetics (PK) of AT-1501
Exploratory- Pharmacokinetic Parameters- Vdss | T=0 (pre infusion), 1 (end of infusion), 2, 4, 8, 12, 24 and 48 hrs.
  Pharmacokinetics (PK) of AT-1501
Exploratory- Pharmacokinetic Parameters- (t1/2) | T=0 (pre infusion), 1 (end of infusion), 2, 4, 8, 12, 24 and 48 hrs.
  Pharmacokinetics (PK) of AT-1501

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Bornstein, MD, Study Chair — Eledon Pharmaceuticals
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada